CLINICAL TRIAL: NCT04723940
Title: Oral vs Intravenous Antibiotics for Treatment of Periprosthetic Joint Infection
Brief Title: Or v IV Antibiotics for Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JPAR 20D.1085
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Joint Infection
MeSH Terms: interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Cefadroxil; Clindamycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Antibiotics (Active Comparator): Participant will receive 6 weeks of oral antibiotic therapy to treat their infection. The type of antibiotic given will be at the discretion of the infectious disease doctor.
  Interventions: Drug: Bactrim; Drug: Cefadroxil; Drug: Doxycycline Hcl; Drug: Clindamycin
- Intravenous Antibiotics (Active Comparator): Participant will receive 6 weeks of intravenous (IV) antibiotic therapy to treat their infection. The type of antibiotic given will be at the discretion of the infectious disease doctor.
  Interventions: Drug: Bactrim; Drug: Cefadroxil; Drug: Doxycycline Hcl; Drug: Clindamycin

INTERVENTIONS:
Drug: Bactrim — Bactrim will be given for 6 weeks to treat joint infection
Drug: Cefadroxil — Cefadroxil will be given for 6 weeks to treat joint infection
Drug: Doxycycline Hcl — Doxycycline HCl will given for 6 weeks to treat joint infection
Drug: Clindamycin — Clindamycin will given for 6 weeks to treat joint infection

SUMMARY:
Management of periprosthetic joint infection (PJI) commonly includes 6 weeks of intravenous (IV) antibiotics after surgical treatment. However, there is little evidence to suggest that oral (PO) therapy results in worse outcomes. This study aims to determine whether or not PO antibiotics are non-inferior to IV antibiotics in treating PJI. The study is a multicenter, parallel-group, randomized (1 : 1), open-label, non-inferiority trial. The non-inferiority margin will be set at 10%. Adults with a clinical diagnosis of PJI according to the International Consensus Meeting (ICM) criteria who would ordinarily receive at least 6 weeks of antibiotics and have received ≤ 7 days of IV therapy from surgery will be included. A total of 308 participants will be centrally computer-randomized to PO or IV antibiotics to complete the first 6 weeks of therapy. Follow-on PO therapy will be permitted in either arm. The primary outcome is the proportion of participants experiencing treatment failure within 1 year. An associated cost-effectiveness evaluation including complications, resource utilization and quality-of-life data will be performed.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* willing and able to give informed consent
* primary THA or TKA diagnosed with PJI based on International Consensus Meeting criteria

  1. A sinus communicating with the prosthesis OR
  2. Two positive cultures obtained from the prosthesis OR
  3. 3 of 5 criteria:
* Elevated ESR (>30mm/hr) and CRP (>10mg/L)
* Elevated synovial leukocyte count (>3000 cells/µL) or change of ++ on leukocyte esterase strip
* Elevated synovial neutrophil percentage (>80%)
* One positive culture
* Positive histological analysis of periprosthetic tissue (>5 neutrophils per high power field in 5 high power fields x400)
* PJI treated by debridement and implant retention, or excision of the prosthetic joint (with or without planned reimplantation)
* received ≤ 7 days of IV therapy after an appropriate surgical intervention

Exclusion Criteria:

* Previously treated for native septic arthritis or PJI in the same joint
* S. aureus bacteremia on presentation or within the previous month
* clinical, histological or microbiological evidence of mycobacterial, fungal or parasitic etiology of the infection
* any other concomitant infection that, in the opinion of the clinician responsible for the patient, requires a prolonged course of IV antibiotic therapy (e.g. bacterial endocarditis, mediastinal infection, central nervous system infection)
* septic shock or systemic features that, in the opinion of the clinician responsible for the patient, requires a course of IV antibiotic therapy (the patient could be re-evaluated if these features resolved)
* an infection for which there are no suitable antibiotic choices to permit randomization between the two arms of the trial (e.g. when organisms are only sensitive to IV antibiotics or PO antibiotics)
* unlikely to comply with trial requirements following randomization in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2023-01-25 (Estimated); Study Completion 2023-01-25 (Estimated)

PRIMARY OUTCOMES:
Rate of Postoperative Infections | 2 years
  The investigator will measure the incidence of postoperative infections in participants treated with oral antibiotics versus those treated with intravenous antibiotics

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States